CLINICAL TRIAL: NCT07147179
Title: Pilot Trial of Short Course Radiotherapy for Primary or Secondary CNS Malignancies
Brief Title: Short Course Radiotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 27924; 858464 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2025-08-27; First posted 2025-08-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Central Nervous System Cancer
Keywords: Short Course; Radiotherapy
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Short Course Radiotherapy (Experimental): Short-course radiation therapy in pediatric patients with incurable central nervous system malignancies
  Interventions: Radiation: Short Course Radiotherapy

INTERVENTIONS:
Radiation: Short Course Radiotherapy — Participants will receive a shorter course of radiation therapy across 5 days (20 Gray in 5 fractions).

SUMMARY:
This is a single arm prospective pilot trial determining the safety of short-course radiation therapy in pediatric patients with incurable central nervous system malignancies.

DETAILED DESCRIPTION:
Participants will receive a shorter course of radiation therapy across 5 days (20 Gray in 5 fractions) in contrast to the standard treatment of two weeks or more of daily treatments (up to 3 Gray per day). This research study is being conducted to see if delivering a shorter course of radiation therapy is safe and helps quality of life so that it may reduce the required duration of palliative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 21 years or below
* Lansky performance status >= 40
* Has a diagnosis of an incurable malignancy that:

  * Originates outside the brain but is metastatic to 1 or more sites within the brain, or originates and recurs within the brain. For this diagnosis to be confirmed, there must be multidisciplinary review of up to date imaging at a pediatric tumor board with unanimous consensus of intracranial relapse or metastasis. If the consensus is not unanimous, short-interval repeat imaging with subsequent unanimous consensus would be required in order for this eligibility criteria to be met
  * Has at least 1 targetable intracranial lesion as seen on imaging
  * Has a multidisciplinary consensus recommendation for palliative intent radiation
* Consents to the study or has caregiver who is able to provide signed and dated informed consent. For subjects under the age of 18, a signed and dated assent form as able.
* Patients who had prior radiation in planned treatment area are also eligible to enter the trial
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Radiotherapy for curative intent
* Serious uncontrolled systemic or psychiatric disorders that would interfere with participation in the protocol
* Being planned for proton radiation

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety of Short Course Radiotherapy | 1 year
  The ability to complete short-course radiotherapy without grade 3 or higher adverse events (AE) that are possibly, probably, or definitely related to radiotherapy during the study period
  Any individual grade 3 or higher AE that is reported during the study period and deemed possibly, probably, or definitely related to short course radiotherapy will automatically prevent the study from meeting its primary endpoint.

SECONDARY OUTCOMES:
Pediatric Quality of Life after Short Course Radiotherapy | 1 year
  Trends in composite scores from validated pediatric quality of life instruments, including PedsQLTM (Pediatric Quality of Life Inventory, Children's Hospital and Health Center, San Diego, California), for patients ages 0-18 years, administered at each prespecified time period
Adolescent Quality of Life after Short Course Radiotherapy | 1 year
  Trends in composite scores from validated adolescent quality of life instruments, including FACT-Br (Functional Assessment of Cancer Therapy-Brain) for patients 18-21 years, administered at each prespecified time period
Overall Survival after Short Course Radiotherapy | 1 year
  Time (in weeks) from the last day of radiotherapy to death from any cause
Steroid Usage | 1 year
  A binary endpoint whereby total daily steroid requirement is either increased or not increased compared to the immediately preceding study time point
  Radiotherapy may result in swelling leading to an increase in neurological symptoms/signs. We will use need for increase in steroid dosing as a surrogate for global neurological function.

OTHER OUTCOMES:
Rates of brain necrosis | 1 year
  Rates of radiographic and/or pathologic radionecrosis as determined by brain MRI or autopsy findings (if clinically available)

CONTACTS AND LOCATIONS:
Overall Officials: Michael LaRiviere, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No